CLINICAL TRIAL: NCT01090297
Title: CPAP Treatment : Fixed Versus Auto-adjusting Mode Impact on Clinical Blood Arterial Pressure. Randomised, Controlled and Double Blinded Trial in SAOS Patients
Brief Title: Continuous Positive Airway Pressure (CPAP) Mode Impact on Clinical Blood Arterial Pressure
Acronym: AgirSASadom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGIR à Dom (Other)
Responsible Party: Jean Louis PEPIN, CHU de Grenoble
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGIR-01
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2011-04

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; Blood pressure; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed pressure (Active Comparator)
  Interventions: Device: S8 Spirit 2; Device: Somnosmart 2; Device: Remstar Auto
- Auto-adjusting pressure (Active Comparator)
  Interventions: Device: S8 Spirit 2; Device: Somnosmart 2; Device: Remstar Auto

INTERVENTIONS:
Device: S8 Spirit 2 — 3 types of Continuous Positive Airway Pressure (CPAP) device: S8 Spirit 2, Somnosmart 2, Remstar Auto.
  These 3 types of CPAP can be set in both mode of pressure.
Device: Somnosmart 2 — 3 types of Continuous Positive Airway Pressure (CPAP) device: S8 Spirit 2, Somnosmart 2, Remstar Auto.
  These 3 types of CPAP can be set in both mode of pressure.
Device: Remstar Auto — 3 types of Continuous Positive Airway Pressure (CPAP) device: S8 Spirit 2, Somnosmart 2, Remstar Auto.
  These 3 types of CPAP can be set in both mode of pressure.

SUMMARY:
Background: Continuous positive airway pressure (CPAP) is the first line therapy for obstructive sleep apnea syndrome (OSAS). Two positive airway pressure (PAP) modalities can be used: Fixed pressure, in which the effective pressure is set and kept constant all night, and auto CPAP devices where the positive pressure changes during the night depend on patient's requirements.

Hypothesis: Pressure variations associated with autoCPAP functioning can lead to sleep fragmentation and alterations in sleep structure. This can limit blood pressure dipping during sleep and then impact clinical blood pressure reduction.

Main objective: To compare in a randomized controlled trial 4 months clinical blood pressure (BP) evolution depending on CPAP mode: fixed pressure versus autoCPAP. Secondary outcomes: Evolution of arterial stiffness, biological parameters, quality of life and symptoms.

Methods: Patients will be randomised depending on CPAP mode. Baseline and 4 months evaluation will include: 24-h ambulatory blood pressure monitoring, clinical BP measurements and carotid-to-femoral pulse wave velocity (PWV). Patients will also complete quality of life and symptoms questionnaires.

2 interim analysis will be carried out when 150 and 220 patients respectively will have completed the study. The Peto's method will be used to correct the p-values.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* patients who gave written informed consent
* patients who subscribed a social insurance
* SAOS patients who need CPAP treatment.

Exclusion Criteria:

* cardiac failure known and treated
* central Apnea syndrome
* patients who stopped CPAP treatment in the previous year
* pregnant women
* patients under guardianship
* imprisoned patients, patients in hospital
* patients included in an other clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Clinical blood pressure | Before treatment, 4 months after treatment

SECONDARY OUTCOMES:
Pulse Wave Velocity | Before treatment, 4 months after treatment
24 hours Blood Pressure measure | Before treatment, after 4 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- AGIR à Dom, Meylan, France

REFERENCES:
- [Derived] Pepin JL, Tamisier R, Baguet JP, Lepaulle B, Arbib F, Arnol N, Timsit JF, Levy P. Fixed-pressure CPAP versus auto-adjusting CPAP: comparison of efficacy on blood pressure in obstructive sleep apnoea, a randomised clinical trial. Thorax. 2016 Aug;71(8):726-33. doi: 10.1136/thoraxjnl-2015-207700. Epub 2016 Apr 18. PMID 27091542